CLINICAL TRIAL: NCT04074291
Title: Cross Cultural Validation of the Italian Version of the Bt-DUX: A Subjective Measure of Health Related Quality of Life in Patients Who Underwent Surgery for Lower Extremity Malignant Bone Tumour
Brief Title: Cross Cultural Validation of the Italian Version of the Bt-DUX
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 441/2019/Oss/IOR
Record Dates: First submitted 2019-07-17; First posted 2019-08-30 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-02

CONDITIONS: Quality of Life; Bone Neoplasm
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the presented study is to translate the English Bt-DUX (Bt-DUX-Eng) questionnaire into the Italian language and then examine the validity of the Italian version of the Bt-DUX (Bt-DUX-It).

DETAILED DESCRIPTION:
Validation of the Italian Bt-DUX:

Cross sectional study among patients of the Istituto Ortopedico Rizzoli, Bologna, Italy, will carry out. All patients who underwent a surgical intervention due to a malignant bone tumour in the leg will be identified through hospital records and a survey consisting of different QoL questionnaires will be executed:

Bt-DUX, EORTC QLQ C-30, The Toronto Extremity Salvage Score (TESS).

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they're aged between 15 and 25 years at the time of the selection, if the time since surgery is ranged between 12 and 60 months, if the malignant bone tumour (osteosarcoma or Ewing's sarcoma) was located around the hip or the knee and the surgical intervention consisted of limb sparing or ablative surgery.

Exclusion Criteria:

* Patients will be excluded if other medical conditions limit their physical activities.

Ages: 15 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients who underwent a surgical intervention due to a malignant bone tumour in the leg will be identified through hospital records of Istituto Ortopedico Rizzoli.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Bt-DUX.it | Between 12 and 60 months after the surgery
  The disease specific Bt-DUX relates to the patient's subjective feeling about a specific aspect, using abstract faces (smiley's) as answer categories. The expressions from very happy to sad (score 1-5) form a five-point Likert scale. The Bt-DUX consists of 20 questions which cover the domains social, emotional, cosmetical and physical functioning. Single item scores were recoded and computed into raw total and domain scores. These raw scores were converted into total and domain scores, ranging from 0-100, with the highest scores indicating better QoL .

SECONDARY OUTCOMES:
The Toronto Extremity Salvage Score (TESS) | Between 12 and 60 months after the surgery
  The Toronto Extremity Salvage Score (TESS), a validated and reliable disease-specific measure developed to evaluate physical disability in patients treated for extremity sarcoma. The self-administered questionnaire includes 30 items on activity limitations in daily life, such as restrictions in body movement, mobility, self-care and performance of daily tasks and routine. The degree of physical disability is rated from 0 (not possible) to 5 (without any problem). The raw score is converted to a score ranged from 0 to 100 points, with higher scores indicating no functional limitations.
EORTC QLQ (Quality of Life Questionnaire) C-30. | Between 12 and 60 months after the surgery
  The 30-item EORTC QLQ-C30 questionnaire is composed of scales that evaluate physical functioning and role functioning, as well as emotional, social, and cognitive functioning and global QOL. Three symptom scales measure fatigue, pain, and emesis, while six single items assess financial impact and physical symptoms such as dyspnoea, sleep disturbance, appetite, diarrhoea, and constipation. The time frame is the past week. The questions are formatted with either yes or no answers, or by using four-answer categories that range from 1, not at all, to 4, very much. The two questions on general health and global QOL are to be answered on a numbered visual-analogue scale from I to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Forni, Study Chair — Isituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Bekkering WP, Vlieland TP, Koopman HM, Schaap GR, Schreuder HW, Beishuizen A, Tissing WJ, Hoogerbrugge PM, Anninga JK, Taminiau AH. The Bt-DUX: development of a subjective measure of health-related quality of life in patients who underwent surgery for lower extremity malignant bone tumor. Pediatr Blood Cancer. 2009 Sep;53(3):348-55. doi: 10.1002/pbc.22078. PMID 19459200
- [Background] Bekkering WP, Billing L, Grimer RJ, Vlieland TP, Koopman HM, Nelissen RG, Taminiau AH. Translation and preliminary validation of the English version of the DUX questionnaire for lower extremity bone tumor patients (Bt-DUX): a disease-specific measure for quality of life. J Surg Oncol. 2013 Mar;107(4):353-9. doi: 10.1002/jso.23218. Epub 2012 Jul 17. PMID 22806913
- [Background] Davis AM, Wright JG, Williams JI, Bombardier C, Griffin A, Bell RS. Development of a measure of physical function for patients with bone and soft tissue sarcoma. Qual Life Res. 1996 Oct;5(5):508-16. doi: 10.1007/BF00540024. PMID 8973131
- [Background] Apolone G, Filiberti A, Cifani S, Ruggiata R, Mosconi P. Evaluation of the EORTC QLQ-C30 questionnaire: a comparison with SF-36 Health Survey in a cohort of Italian long-survival cancer patients. Ann Oncol. 1998 May;9(5):549-57. doi: 10.1023/a:1008264412398. PMID 9653497
- [Background] van Doorn RK, Winkler LM, Zwinderman KH, Mearin ML, Koopman HM. CDDUX: a disease-specific health-related quality-of-life questionnaire for children with celiac disease. J Pediatr Gastroenterol Nutr. 2008 Aug;47(2):147-52. doi: 10.1097/MPG.0b013e31815ef87d. PMID 18664865
- [Background] Vrijmoet-Wiersma CM, Kooloos VM, Koopman HM, Kolk AM, van der Laan I, Grootenhuis MA, Egeler RM. Health-related quality of life, cognitive functioning and behaviour problems in children with Langerhans cell histiocytosis. Pediatr Blood Cancer. 2009 Jan;52(1):116-22. doi: 10.1002/pbc.21740. PMID 18819122
- [Background] Bekkering WP, Vliet Vlieland TP, Koopman HM, Schaap GR, Beishuizen A, Anninga JK, Wolterbeek R, Nelissen RG, Taminiau AH. A prospective study on quality of life and functional outcome in children and adolescents after malignant bone tumor surgery. Pediatr Blood Cancer. 2012 Jun;58(6):978-85. doi: 10.1002/pbc.23328. Epub 2011 Oct 11. PMID 21990185
- [Background] Bekkering WP, Vliet Vlieland TP, Fiocco M, Koopman HM, Schoones JW, Nelissen RG, Taminiau AH. Quality of life, functional ability and physical activity after different surgical interventions for bone cancer of the leg: A systematic review. Surg Oncol. 2012 Jun;21(2):e39-47. doi: 10.1016/j.suronc.2011.09.002. Epub 2011 Oct 4. PMID 21974808
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Koopman HM, Koetsier JA, Taminiau AH, Hijnen KE, Bresters D, Egeler RM. Health-related quality of life and coping strategies of children after treatment of a malignant bone tumor: a 5-year follow-up study. Pediatr Blood Cancer. 2005 Oct 15;45(5):694-9. doi: 10.1002/pbc.20408. PMID 15924359
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752

DOCUMENTS (1):
  • Study Protocol (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT04074291/Prot_000.pdf